CLINICAL TRIAL: NCT01902485
Title: Immediate Initiation of Progestin Contraceptives in First Trimester Medical Abortion: A Randomized Controlled Trial
Brief Title: Study of Immediate Start of Progestin Contraceptives in Medical Abortion
Acronym: Quickstart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1009
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Contraception
Keywords: Contraception; Medical Abortion; Implant; Injectable; Quickstart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quickstart (Active Comparator): Immediate start
  Interventions: Other: Timing of Contraceptive Initiation in Medical Abortion
- Afterstart (Active Comparator): Delayed start
  Interventions: Other: Timing of Contraceptive Initiation in Medical Abortion

INTERVENTIONS:
Other: Timing of Contraceptive Initiation in Medical Abortion

SUMMARY:
This study will compare immediate to post-abortion start of two progestin-based contraceptives (DMPA and etonorgestrel implants) among women having first trimester medical abortion who wish to use that method for post-abortion contraception.

ELIGIBILITY:
Inclusion Criteria:

Women having medical abortion desiring progestin-based contraceptives (injectables or implants)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 937 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Medical Abortion Failure | One month after enrollment
Repeat Pregnancy | 6 months after enrollment

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Planned Parenthood of the Pacific Southwest, Chula Vista, California
  - Planned Parenthood Northern California, Eureka, California
  - Planned Parenthood of Southern New England, Stamford, Connecticut
  - Bayview Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
- Mexico (2):
  - Centro de Salud Beatriz Velasco de Aleman, Mexico City
  - Centro de Salud Santa Catarina, Mexico City

REFERENCES:
- [Derived] Raymond EG, Weaver MA, Louie KS, Tan YL, Bousieguez M, Arangure-Peraza AG, Lugo-Hernandez EM, Sanhueza P, Goldberg AB, Culwell KR, Kaplan C, Memmel L, Sonalkar S, Jamshidi R, Winikoff B. Effects of Depot Medroxyprogesterone Acetate Injection Timing on Medical Abortion Efficacy and Repeat Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2016 Oct;128(4):739-45. doi: 10.1097/AOG.0000000000001627. PMID 27607859
- [Derived] Raymond EG, Weaver MA, Tan YL, Louie KS, Bousieguez M, Lugo-Hernandez EM, Arangure-Peraza AG, Sanhueza P, Kaplan C, Sonalkar S, Goldberg AB, Culwell KR, Memmel L, Jamshidi R, Winikoff B. Effect of Immediate Compared With Delayed Insertion of Etonogestrel Implants on Medical Abortion Efficacy and Repeat Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2016 Feb;127(2):306-12. doi: 10.1097/AOG.0000000000001274. PMID 26942358